CLINICAL TRIAL: NCT01807091
Title: Feasibility of Outpatient Induction Chemotherapy for Adult Patients With Acute Myeloid Leukemia or Advanced Myelodysplastic Syndrome
Brief Title: Outpatient Induction Chemotherapy in Treating Patients With Acute Myeloid Leukemia or Advanced Myelodysplastic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elihu H. Estey, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7910; NCI-2013-00483 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7910 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1000945 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Adult Acute Myeloid Leukemia; Adult Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy) (Experimental): Participants received intensive initial or salvage induction chemotherapy regimens. These regimens would usually be administered in the inpatient setting, however participants received them outpatient. This study did not dictate the choice of induction chemotherapy regimen. The regimen was decided upon by patient and their treating oncologist and clinical care team. The induction chemotherapy regimens administrations spanned 4-7 days.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Receive outpatient induction chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General

SUMMARY:
This pilot clinical trial studies the feasibility of having induction chemotherapy in an outpatient setting. Patients with acute leukemia (AML) or advanced myelodysplastic syndrome (MDS), at least 18 years of age will be examined. Treating eligible patients with induction chemotherapy in an outpatient setting may save in healthcare cost and improve a patients' quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Assess the feasibility of outpatient induction therapy for acute myeloid leukemia (AML) or advanced myelodysplastic syndrome (MDS) by examining whether:

1. > 50% of patients treated as outpatients can complete chemotherapy without being admitted to hospital.
2. < 5% of patients die within 14 days of beginning outpatient chemotherapy.

OUTLINE:

Patients receive outpatient induction chemotherapy.

STATISTICAL CONSIDERATIONS:

The study was monitored to assure that there was not an excess probability of admission to the hospital during receipt of outpatient chemotherapy or death within 14 days of initiating chemotherapy as assessed by Bayesian posterior probabilities using the "predictive probabilities" tool (MD Anderson Cancer Center Department of Statistics).

Stopping earlier would happen under 2 circumstances:

1. Excess probability that patients required admission to hospital during the 4-7 days of outpatient chemotherapy (predictive probability be < 0.10, or 7 patients admitted and 3 not admitted among 10 patients enrolled versus the maximum acceptable rate of 4 patients admitted and 6 not admitted among 10 patients enrolled).
2. Excess probability that patients die during the 14 days after beginning outpatient treatment (predictive probability be >0.90, for example in cases where there are 2 patient deaths within 14 days and less than 5 patients without deaths within 14 days, or in any case where there are 3 patient deaths within 14 days).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent

  * The signed informed consent
  * The benefits/risks of the induction chemotherapy regimen will be reviewed, and a second consent may be necessary if the regimen will be administered according to a separate protocol
* AML (acute promyelocytic leukemia [APL] excepted) or high-risk MDS (10-19% blasts in marrow by morphology or flow cytometry or blood)
* Treatment-related mortality (TRM) score < 9.21 corresponding to a TRM rate of 3% when chemotherapy of similar intensity as proposed here is administered to inpatients
* Blast count =< 10,000
* Fibrinogen > 200
* Afebrile with clear chest imaging and no signs of active viral, bacterial, fungal infection unless determined to be, at the discretion of the investigator, not clinically significant in the context of this study
* Adequate cardiac function as demonstrated by left ventricular ejection fraction (LVEF) of 45% or greater, by multiple gated acquisition (MUGA) or echocardiogram; no ongoing cardiac issues such as uncontrolled arrhythmias or unstable angina or congestive heart failure
* Patient must have an outpatient caregiver available
* Patient must live within 30 minutes of the treating physician's office during outpatient treatment
* Patient must be willing to return to the treating physician's office for outpatient follow-up once outpatient treatment is completed
* Logistical requirements:

  * Space available in infusion room
  * Outpatient infusion pump available if continuous infusion required
  * Case discussed with infusion room nursing staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Becker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Eli Estey, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (9):
- United States (9):
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Group Health Cooperative, Redmond, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Multicare Health System, Tacoma, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy)
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 53 [19 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Treatment Related Mortality (TRM) score [Median (Full Range); unit: units on a scale (0-100)] — Our institution defines TRM as death within 28 days from initiation of chemotherapy based on the observation that the risk of death declines once 4 weeks has elapsed from treatment start. A calculation is used to predict TRM using patient's age, performance status, if they have secondary AML, albumin, creatinine, platelet count, white blood cell count, and peripheral blood blast percentage. The higher the TRM score, the higher the risk of TRM. Calculator and table of relationship between TRM score and TRM probability found here: https://cstaging.fhcrc-research.org/TRM/Default.aspx
  units on a scale (0-100) | 1.6 [0.0 to 8.0]
Disease [Count of Participants; unit: Participants]
  AML | 15
  MDS (EB-2) | 2
Disease status [Count of Participants; unit: Participants]
  Newly diagnosed | 8
  Relapsed or refractory | 9
Induction chemotherapy regimen [Count of Participants; unit: Participants]
  Idarubicin, cytarabine, pravastatin (IAP) | 2
  Cladribine, cytarabine, mitoxantrone, granulocyte colony-stimulating factor (GCLAM) | 7
  Decitabine, cladribine, cytarabine, mitoxantrone, granulocyte colony-stimulating factor (D-GCLAM) | 2
  Clofarabine, cytarabine, granulocyte colony-stimulating factor (GCLAC) | 3
  Decitabine, mitoxantrone, etoposide, cytarabine (D-MEC) | 3
Number of days of predetermined treatment [Median (Full Range); unit: Days of predetermined treatment] — This measure describes the median length (in number of days) the outpatient induction chemotherapy regimen would be administered and was scheduled for. Induction chemotherapy regimen was decided upon by subject, their treating oncologist and clinical care team.
  Days of predetermined treatment | 5 [4 to 5]
Year enrolled [Count of Participants; unit: Participants]
  2010-2013 | 1
  2014-2018 | 16
Hematocrit on day 1 [Median (Full Range); unit: Percentage of red blood cells in blood] | 28 [23 to 40]
Platelet count on day 1 [Median (Full Range); unit: 10 x 10^9 cells/L] | 71 [12 to 1108]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Hospital Admission During Outpatient Induction Chemotherapy
Description: Feasibility for this study objective would be considered a "success" if >50% of patients treated as outpatients can complete chemotherapy without being admitted to hospital.
Time Frame: During the 4-7 days of outpatient induction chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 17
Participants
  Admitted during induction chemotherapy period | 3
  Not admitted during induction chemotherapy period | 14

2. Primary Outcome: Death Within 14 Days of Initiating Outpatient Induction Chemotherapy
Description: Feasibility for this study objective would be considered a "success" if <5% of patients die within 14 days of beginning outpatient chemotherapy.
Time Frame: During the 14 days after beginning outpatient induction treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 17
Participants | 0

ADVERSE EVENTS:
Time Frame: From the start of outpatient chemotherapy through day 14 after starting outpatient chemotherapy.
Description: Only the following adverse events were recorded:
  1. Reasons for hospitalization during planned outpatient administration of chemotherapy
  2. Causes of any deaths that occur within 14 days of start of outpatient chemotherapy
  Other adverse events were not monitored/assessed.
Arm/Group | Treatment (Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy) (N=17)
Neutropenic fever (Infections and infestations) | 2 (2)
Mucositis (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Slow accrual was due to initial limitation of enrollment to younger patients receiving initial induction. It was expanded to include older patients, including those receiving salvage induction. The ability to give outpatient induction was often logistically limited. Because of these issues, only 17 patients were treated and it is likely there was significant selection bias, complicating interpretation of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT01807091/Prot_SAP_000.pdf